CLINICAL TRIAL: NCT04282486
Title: Medication Exposure in Older Patients (AGEd > 65 Years) With Constitutional HEMORRHagic Disease (Haemophilia or Willebrand Disease).
Brief Title: Medication Exposure in Older Patients With Constitutional Hemorrhagic Disease
Acronym: M-HEMORRH'AGE
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL20_0086
Record Dates: First submitted 2020-02-21; First posted 2020-02-24 (Actual); Last update posted 2021-07-13 (Actual); Status verified 2021-07

CONDITIONS: Hemophilia
Keywords: Willebrand disease
MeSH Terms: conditions — Hemophilia A | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Telephone interview — Primary objective: potentially inappropriate medication prevalence
  Secondary objective:
  Number and type of medication Polypharmacy prevalence Medication regimen complexity using Medication Regimen Complexity Index Anticholinergic and sedative exposure using Drug Burden Index
  A telephone interview will be conducted with patients in order to collect medication data from medical prescriptions.

SUMMARY:
The improvements observed in the care of patients with hemophilia or Willebrand disease have led to an increase in their life expectancy, which today approaches that of the general population. This increase in life expectancy leads in these patients to the development of comorbidities related to aging (cardiovascular and neurological diseases, cancers and kidney diseases) (e.g "Franchini & Mannuccio", BJH, 2009). The care of these comorbidities represents a new challenge for the medical teams. Toward multiple comorbidities, polypharmacy is often associated.

Many studies about medication exposure and management in older patients were published but no study was conducted to explore the medication management of older patients with hemophilia or Willebrand disease.

ELIGIBILITY:
Inclusion Criteria:

* Community-dwelling patients over 65 years with hemophilia (A or B)
* Community-dwelling patients over 65 years with Willebrand disease (Type1, 2 and 3, rate <30%)

Exclusion Criteria:

* Patients without phone number
* Non French speaking patients

Max Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Elderly patients with hemophilia or Willebrand's disease (over 65) will have a telephone interview in order to collect medication data from medical prescriptions.
Sampling Method: Non-Probability Sample
Enrollment: 142 (Actual)
Dates: Start 2020-07-22 (Actual); Primary Completion 2021-01-29 (Actual); Study Completion 2021-01-29 (Actual)

PRIMARY OUTCOMES:
Potentially inappropriate medication (PIM) prevalence using EU-(7) PIM list. | At inclusion
  A telephone interview will be conducted with patients in order to collect medication data from medical prescriptions. After collection of data for all patients, the research of PIM was conducted.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital des Charpennes, Institut du Vieillissement, Villeurbanne, France